CLINICAL TRIAL: NCT01229657
Title: Study of the Anatomic and Visual Outcomes in Patients With Initially Closed Macular Holes After Vitreoretinal Surgery
Brief Title: Evaluation of Anatomic and Visual Outcomes of Initially Closed Macular Holes
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Shaochong Zhang, Zhongshan Ophthalmic Center, Sun Yat-sen University
Other Study IDs: SunYat-senU; 2008B030301306 (Other Grant/Funding Number: Science and Technology Projects of Guangdong Province); 2007B031302007 (Other Grant/Funding Number: Science and Technology Projects of Guangdong Province)
Record Dates: First submitted 2010-10-27; First posted 2010-10-28 (Estimated); Last update posted 2010-10-28 (Estimated); Status verified 2010-10

CONDITIONS: Macular Holes
Keywords: Reopening of macular hole;; Visual acuity;; Phacoemulsification cataract surgery;; Vitrectomy
MeSH Terms: conditions — Retinal Perforations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To evaluate the anatomic and visual outcomes in patients with initially closed macular holes after vitreoretinal surgery and with one to seven years of follow-up.

DETAILED DESCRIPTION:
In recent years, peeling of the internal limiting membrane (ILM) has been used as a supplementary treatment to reducing the tangential tractional forces and inducing hole closure in macular hole surgery, and thus the anatomic success rate has increased to over 90%. However, despite these high rates of surgical success, the reopening of initially closed macular holes has also been observed from the first month to several years following surgery. Because about 45% to 95% of phakic patients frequently develop a progressive nuclear sclerosis cataract after macular hole surgery and require combined or subsequent cataract extraction to improve visual acuity, cataract extraction has become a potential factor in causing macular hole reopening, although this is still under debate. The purpose of this study is to describe the long-term anatomic and visual outcomes in patients who had initial anatomic success with macular hole surgery and who had postoperative follow-up of one or more years. All patient's charts were reviewed for age, macular hole stage (using the Gass classification), macular hole duration, epiretinal membrane of macula presence, ILM peeling, preoperative and postoperative visual acuity, rate of macular hole reopening, cataract extraction, and length of follow-up after vitrectomy.

ELIGIBILITY:
Inclusion Criteria:

* successful closure of a macular hole after initial vitreoretinal surgery
* a follow-up of at least one year

Exclusion Criteria:

* post-traumatic holes,
* myopic macular holes,
* macular holes associated with a rhegmatogenous retinal detachment,
* eyes with silicone oil tamponade.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with initially closed macular holes after vitreoretinal surgery and with one to seven years of follow-up
Sampling Method: Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2010-03; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shaochong Zhang, MD, Study Chair — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China